CLINICAL TRIAL: NCT06182189
Title: Studio Osservazionale Sulla qualità di Vita di Pazienti Affetti da IPB in Terapia Medica e/o Sottoposti a Intervento Chirurgico
Brief Title: Protocollo N 2014 - Benign Prostatic Hyperplasia
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: 2014 - IPB
Record Dates: First submitted 2023-11-21; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; urology
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a benign prostatic hyperplasia condition: Patients with a benign prostatic hyperplasia condition
  Interventions: Other: Observation of patients with a benign prostatic hyperplasia condition

INTERVENTIONS:
Other: Observation of patients with a benign prostatic hyperplasia condition — Observation of patients with a benign prostatic hyperplasia condition who have undergone surgery

SUMMARY:
Prospective observational study on the quality of life of patients with BPH under medical therapy and/or undergoing surgery.

DETAILED DESCRIPTION:
Prospective observational study on the quality of life of patients with BPH under medical therapy and/or undergoing surgery.

Data relating to the clinical conditions (state of the disease, psychological and related to the quality of life) of patients suffering from BPH under medical therapy and/or undergoing surgery will be collected within a specially designed database which will allow us to easily and secure extraction of data used for statistical analyzes in clinical research.

ELIGIBILITY:
Inclusion Criteria:

* subjects suffering from benign prostatic hyperplasia undergoing medical therapy and/or undergoing surgery
* subjects >= 18 years old
* signature of informed consent

Exclusion Criteria:

* subjects < 18 years
* presence of mental or physical disability that may prevent the patient from answering the questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from benign prostatic hyperplasia undergoing medical therapy and/or undergoing surgery
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Medical history | Baseline
  - patient's medical history, past surgical history, family medical history, social history, allergies, medications;
Psycho-behavioural data - male sexual health | Baseline and up to 6 months
  Male sexual health assessed through the Questionnaire for the evaluation of male sexual health" MSHQ(25-item, range: 7 - 80, greater score indicating better function,
Physical examination - Body temperature | Baseline
  Body temperature detection (Celsius degree)
Psycho-behavioural data - erectile function | Baseline and up to 6 months
  Erectile function assessed through the "International Index of Erectile Function" questionnaire IIEF (scoring: 1 - 30 - 6-10: severe; 11-16: Moderate; 17-25: mild; 26-30: absence
Prostatic Symptoms | Baseline and up to 6 months
  Prostatic Symptoms assessed through the IPSS questionnaire, International Prostatic Symptoms Score: , Scoring 0 -7, 0-7 mild symptoms, 8-19 moderate symptoms, 20-35 severe symptoms;
Incontinence Symptoms | Baseline and up to 6 months
  Incontinence Symptoms assessed through the ICIQ - International Consultation of Incontinence Questionnaire, ICIQ-SF has a maximum score of 21; the higher the score, the more severe is the UI, but there is no normal score;
Physical examination - Body temperature pulse rate | Baseline
  Pulse rate detection (beats per minute)
Physical examination - respiration assessment | Baseline
  Respiration rate detection (breaths per minute)
Physical examination - blood pressure | Baseline
  Blood pressure detection (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No